CLINICAL TRIAL: NCT03410693
Title: A Randomized, Open Label, Multicenter Phase 2/3 Study to Evaluate the Efficacy and Safety of Rogaratinib (BAY1163877) Compared to Chemotherapy in Patients With FGFR-positive Locally Advanced or Metastatic Urothelial Carcinoma Who Have Received Prior Platinum-containing Chemotherapy
Brief Title: Study of Rogaratinib (BAY1163877) vs Chemotherapy in Patients With FGFR (Fibroblast Growth Factor Receptor)-Positive Locally Advanced or Metastatic Urothelial Carcinoma
Acronym: FORT-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17403; 2016-004340-11 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Rogaratinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rogaratinib (Experimental): Rogaratinib treatment study arm, comprising
  1. Pre-treatment period, including FGFR testing and screening,
  2. Treatment period, and
  3. Follow-up period, including active follow-up and long-term follow-up. Patients will be considered "on study" during the pre-treatment, treatment and active followup periods. During the long-term follow-up period the patients will be considered "off study".
  Interventions: Drug: Rogaratinib (BAY1163877)
- Chemotherapy (Active Comparator): Chemotherapy treatment study arm, comprising
  1. Pre-treatment period, including FGFR testing and screening,
  2. Treatment period, and
  3. Follow-up period, including active follow-up and long-term follow-up. Patients will be considered "on study" during the pre-treatment, treatment and active followup periods. During the long-term follow-up period the patients will be considered "off study".
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Rogaratinib administered as oral (p.o.) tablets twice daily (b.i.d.) continuously
  Arms: Rogaratinib
Drug: Chemotherapy — Chemotherapy as taxane (docetaxel or paclitaxel) or vinflunine administered through intravenous (i.v.) infusion every 3 weeks (on day 1 of a 21-day cycle) The choice of the chemotherapy is at the discretion of the investigator, taking into consideration the status of the authorization or treatment guidelines in the given country.
  Arms: Chemotherapy

SUMMARY:
This is a randomized, open-label, multicenter Phase 2/3 study to evaluate the efficacy and safety of rogaratinib (BAY 1163877) compared to chemotherapy in patients with FGFR-positive locally advanced or metastatic urothelial carcinoma who have received prior platinum-containing chemotherapy.

The primary objective is to demonstrate the superiority of rogaratinib over chemotherapy in terms of objective response rate (before: overall survivial) of urothelial carcinoma patients with FGFR positive tumors.

At randomization, patients will have locally advanced or metastatic urothelial carcinoma and have received at least one prior platinum-containing chemotherapy regimen. Only patients with FGFR1 or 3 positive tumors can be randomized into the study. Archival tumor tissue is adequate for testing of FGFR1 and 3 mRNA expressions, which will be determined centrally using an RNA in situ hybridization (RNA-ISH) test. Approximately 42 % of UC patients with locally advanced or metastatic UC are identified as FGFR-positive by the RNA-ISH cut-off applied.

ELIGIBILITY:
Inclusion Criteria:

* Existence of archival or fresh biopsy for FGFR testing. Mandatory FGFR testing of patients will be performed prior to start of screening. The timing of the FGFR test is at the discretion of the investigator. Investigators should ensure all patients will be eligible in terms of disease status and lines of treatment.
* Documented urothelial carcinoma (transitional cell carcinoma) including urinary bladder, renal pelvis, ureters, urethra meeting all of the following criteria

  * Histologically confirmed (Patients with mixed histologies are required to have a dominant transitional cell pattern.)
  * Locally advanced (T4, any N; or any T, N 2-3) or metastatic disease (any T, any N and M1). Locally advanced bladder cancer must be unresectable i.e. invading the pelvic or abdominal wall (stage T4b) or presenting with bulky nodal disease (N2-3).
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0 or 1
* Disease progression during or following treatment with at least one platinum-containing regimen (patients should have been treated for at least 2 cycles). In patients who received prior adjuvant/ neoadjuvant platinum-containing chemotherapy, progression had to occur within 12 months of treatment.
* High FGFR1 or 3 mRNA expression levels in archival or fresh tumor biopsy specimen quantified as outlined in the lab manual
* At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) in contrast enhanced (unless contraindicated) CT or MRI

Exclusion Criteria:

* Previous or concurrent cancer except

  * cervical carcinoma in situ
  * treated basal-cell or squamous cell skin carcinoma
  * any cancer curatively treated > 3 years before randomization
  * curatively treated incidental prostate cancer (T1/T2a)
* Ongoing or previous treatment with anti-FGFR directed therapies (e.g. receptor tyrosine kinase inhibitors including rogaratinib or FGFR-specific antibodies) or with taxanes or vinflunine
* More than two prior lines of systemic anti-cancer therapy for urothelial carcinoma given for advanced unresectable/ metastatic disease
* Ongoing or previous anti-cancer treatment within 4 weeks before randomization.
* Unresolved toxicity higher than National Cancer Institute's Common Terminology Criteria for Adverse Events, version 4.03 (CTCAE v.4.03) Grade 1 attributed to any prior therapy/ procedure excluding alopecia, anemia and/ or hypothyroidism
* History or current condition of an uncontrolled cardiovascular disease including any of the following conditions:

  * Congestive heart failure (CHF) NYHA (New York Heart Association) > Class 2
  * Unstable angina (symptoms of angina at rest) or new-onset angina (within last 3 months before randomization)
  * Myocardial infarction (MI) within past 6 months before randomization
  * Unstable cardiac arrhythmias requiring anti-arrhythmic therapy. Patients with arrhythmia under control with anti-arrhythmic therapy such as beta-blockers or digoxin are eligible.
* Arterial or venous thrombotic events or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before randomization
* Current evidence of endocrine alteration of calcium phosphate homeostasis (e.g. parathyroid disorder, history of parathyroidectomy, tumor lysis, tumoral calcinosis, paraneoplastic hypercalcemia)
* Current diagnosis of any retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion
* Any hemorrhage / bleeding event ≥ CTCAE v.4.03 Grade 3 within 4 weeks before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (161):
- United States (16):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - University of Kansas Medical Center, Westwood, Kansas
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Compass Oncology, Tigard, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Bon Secours St. Francis Hospital, Greenville, South Carolina
  - Texas Oncology-Denton South, Denton, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Summit Cancer Center, Spokane, Washington
- Australia (7):
  - Mid North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Monash Medical Centre, Clayton, Victoria
- Austria (4):
  - Landesklinikum Krems, Krems
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Ottakring - Wilhelminenspital, Vienna
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Saint-Pierre, Ottignies
- Canada (3):
  - Princess Margaret Hospital-University Health Network, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - Ottawa Hospital-General Campus, Ottawa
- China (10):
  - FuJian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shengyang, Liaoning
  - Fifth Medical Center, General Hospital of the Chinese People, Beijing
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huadong Hospital, Affiliated to Fudan University, Shanghai
- Czechia (4):
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni Thomayerova Nemocnice, Praha 4 - Krc
  - Bata Hospital, Zlín
- Denmark (3):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Rigshospitalet, Copenhagen
  - Herlev Hospital - Oncology Research Dept., Herlev
- Docrates Klinikka, Helsinki, Finland
- France (11):
  - Hopital Jean Minjoz, Besançon
  - Hôpital Saint André - Bordeaux, Bordeaux
  - Centre de Lutte Contre le Cancer François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret - Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes - Marseille, Marseille
  - Cochin - Paris, Paris
  - Hôpital d'Instruction des Armées Begin, Saint-Mandé
  - Clinique Saint Anne, Strasbourg
  - Centre Médico-Chirurgical Foch, Suresnes
- Germany (3):
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
- Prince of Wales Hospital Hong Kong, Shatin, Hong Kong
- Hungary (3):
  - MH Egeszsegugyi Kozpont, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Ireland (2):
  - Cork University Hospital, Cork
  - AMNCH, Dublin
- Israel (5):
  - Rambam Health Corporation, Haifa
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Clalit Health Services Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (11):
  - IRST Istituto Scientifico Romagnolo per studio e cura tumori, Forlì Cesena, Emilia-Romagna
  - AUSL Modena, Modena, Emilia-Romagna
  - A.O.U. di Modena - Policlinico, Modena, Emilia-Romagna
  - A.O. San Camillo-Forlanini, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - IRCCS Istituto Europeo di Oncologia s.r.l. (IEO), Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - A.O.U. San Luigi Gonzaga, Turin, Piedmont
  - A.O.U. Pisana, Pisa, Tuscany
  - A.O.U.I. Verona, Verona, Veneto
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Gunma University Hospital, Maebashi, Gunma
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Akita University Hospital, Akita
  - Kyushu University Hospital, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - Niigata University Medical and Dental Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Toyama University Hospital, Toyama
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Poland (6):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Przychodnia Lekarska KOMED, Konin
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Uniwersytecki Szpital Kliniczny UM we Wroclawiu, Wroclaw
- Portugal (5):
  - Hospital Beatriz Angelo, Loures, Lisbon District
  - IPO Coimbra, Coimbra
  - Hospital CUF Infante Santo, Lisbon
  - CHULN - Hospital Santa Maria, Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
- Russia (5):
  - Krasnoyarsk Regional Clinical Oncology Dispensary, Krasnoyarsk
  - Moscow Scient. Res. Institute of Oncology n.a P.A. Hertzen, Moscow
  - Volga District Med Center FMBA, Nizhny Novgorod
  - Clinical Oncological Dispensary of Omsk Region, Omsk
  - Bashkir State Medical University, Ufa
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
- Slovakia (3):
  - Narodny onkologicky ustav, Bratislava
  - UROEXAM, spol. s r.o., Nitra
  - POKO Poprad s.r.o., Poprad
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Son Espases, Palma de Mallorca, Illes Baleares
  - Hospital del Mar, Barcelona
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Reina Sofía, Córdoba
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Instituto Valenciano de Oncología, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Södersjukhuset, Stockholm
  - Karolinska Institutet, Stockholm
- Switzerland (3):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- United Kingdom (2):
  - Clatterbridge Centre for Oncology, Bebington, Merseyside
  - Royal Marsden Hospital (London), London

REFERENCES:
- [Derived] Sternberg CN, Petrylak DP, Bellmunt J, Nishiyama H, Necchi A, Gurney H, Lee JL, van der Heijden MS, Rosenbaum E, Penel N, Pang ST, Li JR, Garcia Del Muro X, Joly F, Papai Z, Bao W, Ellinghaus P, Lu C, Sierecki M, Coppieters S, Nakajima K, Ishida TC, Quinn DI. FORT-1: Phase II/III Study of Rogaratinib Versus Chemotherapy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma Selected Based on FGFR1/3 mRNA Expression. J Clin Oncol. 2023 Jan 20;41(3):629-639. doi: 10.1200/JCO.21.02303. Epub 2022 Oct 14. PMID 36240478
- [Derived] Grunewald S, Politz O, Bender S, Heroult M, Lustig K, Thuss U, Kneip C, Kopitz C, Zopf D, Collin MP, Boemer U, Ince S, Ellinghaus P, Mumberg D, Hess-Stumpp H, Ziegelbauer K. Rogaratinib: A potent and selective pan-FGFR inhibitor with broad antitumor activity in FGFR-overexpressing preclinical cancer models. Int J Cancer. 2019 Sep 1;145(5):1346-1357. doi: 10.1002/ijc.32224. Epub 2019 Mar 13. PMID 30807645
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants at 111centers in 28 countries from 31 MAY 2018 (first participant first visit) to 27 OCT 2020 (last participant last visit).
Pre-assignment Details: A total of 718 participants signed the informed consent for prescreening, of which 256 participants completed the prescreening, while 462 participants discontinued the prescreening. The discontinuations were due to screening failure (322), other reasons (98), withdrawal by the participant (22), and death (20).
Groups:
- Rogaratinib (BAY1163877)_Overall Population: Participants who were randomized to this group following a 1:1 ratio received rogaratinib 600 mg orally twice a day (b.i.d.) continuously, during a 21-day treatment cycle.
- Chemotherapy_Overall Population: Participants who were randomized to this group following a 1:1 ratio received chemotherapy (docetaxel, paclitaxel or vinflunine) at the discretion of the investigator, as intravenous (i.v.) infusion once every three weeks (on day 1 of a 21-day cycle).
Period: Overall Study
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population
Started | 87 | 88
Started Treatment | 86 | 82
Active Follow-up Performed | 61 | 56
Entered Long Term Follow-up | 56 | 69
Completed (Completed treatment, participants who discontinued treatment could enter follow-up.) | 0 (Completed treatment) | 0 (Completed treatment)
Not Completed | 87 | 88
Not completed — Disc trt: Withdrawal by participant | 6 | 4
Not completed — Disc trt: Lost to follow up | 0 | 1
Not completed — Disc trt: radiological progression | 58 | 50
Not completed — Disc trt: Other | 1 | 0
Not completed — Study drug never administered | 1 | 6
Not completed — Discontinued (disc) treatment (trt): Death | 6 | 4
Not completed — Disc trt: Adverse Event (AE) | 13 | 9
Not completed — Disc trt: Physician decision | 0 | 5
Not completed — Disc trt: clinical progression | 1 | 5
Not completed — Disc trt:AE not asso. w/ clinical disease progress | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.3) | 66.4 (10.3) | 67.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 70 | 145
  Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 76 | 78 | 154
  Unknown or Not Reported | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 23 | 25 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 55 | 55 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
Cancer Category [Count of Participants; unit: Participants]
  Location of primary cancer: bladder | 56 | 45 | 101
  Location of primary cancer: Ureter | 17 | 14 | 31
  Location of primary cancer: Renal pelvis | 12 | 28 | 40
  Location of primary cancer: Proximal urethra | 2 | 1 | 3
Cancer stage at study entry [Count of Participants; unit: Participants] — Higher value/letter correlates to advanced stages of the malignancy. IIIA: The tumor has grown into the perivesical tissue or has spread to the prostate, uterus, or vagina, but has not spread to the lymph nodes or other organs, or cancer has spread to a single regional lymph node; IIIB: the tumor has spread to 2 or more regional lymph nodes or the common iliac lymph nodes; IVA: The cancer has spread to the pelvic wall or the abdominal wall but not to other parts of the body, or has spread to lymph nodes located outside of the pelvis; IVB: the tumor has spread to other parts of the body.
  Participants
    Stage III B | 1 | 3 | 4
    Stage IV | 5 | 12 | 17
    Stage IV A | 13 | 24 | 37
    Stage IV B | 67 | 48 | 115
    Unknown | 1 | 1 | 2
PIK3CA and/or RAS activating mutations [Count of Participants; unit: Participants] — PIK3CA: Phosphoinositide 3 kinase, catalytic subunit alpha isoform RAS: Rat sarcoma
  Participants
    Absent | 65 | 69 | 134
    Present | 10 | 10 | 20
    Unknown | 12 | 9 | 21
FGFR expression from Targos [Count of Participants; unit: Participants] — FGFR: Fibroblast growth factor receptor
  Participants
    Negative | 13 | 14 | 27
    Positive | 69 | 69 | 138
    Not assessed | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - Central Assessment
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR). participants for whom overall best response is not CR or PR, as well as participants without any post-baseline tumor assessment will be considered non-responders.
Time Frame: From start of treatment up to end of active follow-up, approximately 29 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rogaratinib_WT Population: Rogaratinib arm, wild type population
- Chemotherapy_WT Population: Chemotherapy group, wild type population
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population | Rogaratinib_WT Population | Chemotherapy_WT Population
Number analyzed (Participants) | 87 | 88 | 62 | 63
percentage of participants | 19.5 [11.8 to 29.4] | 21.6 [13.5 to 31.6] | 19.4 [10.4 to 31.4] | 23.8 [14.0 to 36.2]
Statistical Analysis 1: Comparison: Rogaratinib (BAY1163877)_Overall Population vs Chemotherapy_Overall Population; Test type: Superiority; p = 0.6991, Fisher Exact; ORR difference (R-C) = -2.1, 95% CI 2-sided [-14.0 to 9.9]
Statistical Analysis 2: Comparison: Rogaratinib_WT Population vs Chemotherapy_WT Population; Test type: Superiority; p = 0.7944, Fisher Exact; ORR difference (R - C) = -4.5, 95% CI 2-sided [-18.9 to 9.9]

2. Secondary Outcome: Disease-control Rate (DCR) - Central Assessment
Description: DCR was defined as the percentage of participants whose overall best response was not a progressive disease (i.e., CR, PR, stable disease [SD] or Non CR/Non PD).
Time Frame: From start of treatment till end of active follow-up, approximately 29 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population | Rogaratinib_WT Population | Chemotherapy_WT Population
Number analyzed (Participants) | 87 | 88 | 62 | 63
percentage of participants | 50.6 [39.6 to 61.5] | 55.7 [44.7 to 66.3] | 53.2 [40.1 to 66.0] | 63.5 [50.4 to 75.3]
Statistical Analysis 1: Comparison: Rogaratinib (BAY1163877)_Overall Population vs Chemotherapy_Overall Population; Test type: Superiority; p = 0.7962, Fisher Exact; DCR difference (R-C) = -5.1, 95% CI 2-sided [-19.9 to 9.7]
Statistical Analysis 2: Comparison: Rogaratinib_WT Population vs Chemotherapy_WT Population; Test type: Superiority; p = 0.9109, Fisher Exact; DCR difference (R-C) = -10.3, 95% CI 2-sided [-27.5 to 6.9]

3. Secondary Outcome: Progression-free Survival (PFS) - Central Assessment
Description: Progression free survival (PFS) was defined as the time (days) from randomization to date of first observed disease progression (radiological or clinical assessment or both) or death due to any cause (if death occurred before progression was documented).
Time Frame: From start of treatment till end of active follow-up, approximately 29 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population | Rogaratinib_WT Population | Chemotherapy_WT Population
Number analyzed (Participants) | 87 | 88 | 62 | 63
months | 2.7 [1.6 to 4.6] | 3.2 [2.7 to 4.4] | 2.8 [2.6 to 5.1] | 4.0 [2.8 to 6.1]
Statistical Analysis 1: Comparison: Rogaratinib (BAY1163877)_Overall Population vs Chemotherapy_Overall Population; Test type: Superiority; p = 0.8672, Log Rank; Hazard Ratio (HR) = 1.226, 95% CI 2-sided [0.853 to 1.762]
Statistical Analysis 2: Comparison: Rogaratinib_WT Population vs Chemotherapy_WT Population; Test type: Superiority; p = 0.9171, Log Rank; Hazard Ratio (HR) = 1.341, 95% CI 2-sided [0.880 to 2.043]

4. Secondary Outcome: Duration of Response (DOR) - Central Assessment
Description: DOR (for patients with PR and CR only) was defined as the time from the first documented objective response of PR or CR, whichever was noted earlier, to disease progression (including symptomatic deterioration) or death, whichever was earlier
Time Frame: From start of treatment till end of active follow-up, approximately 29 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rogaratinib (BAY1163877)_Overall Population | Chemotherapy_Overall Population | Rogaratinib_WT Population | Chemotherapy_WT Population
Number analyzed (Participants) | 87 | 88 | 62 | 63
months | 4.9 [2.2 to 7.0] | 5.8 [3.5 to 7.7] | 5.1 [1.5 to 9.2] | 7.0 [2.7 to 8.4]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: A treatment-emergent event was defined as any event arising or worsening after the start of study drug administration until 30 days after the last administration of study treatment
Time Frame: From start of treatment up to 30 days after the last administration of study treatment, approximately 29 months
Measure: Count of Participants; unit: Participants
Groups:
- Rogaratinib (BAY1163877): Participants who were randomized to this group following a 1:1 ratio received rogaratinib 600 mg orally twice a day (b.i.d.) continuously, during a 21-day treatment cycle.
- Chemotherapy: Participants who were randomized to this group following a 1:1 ratio received chemotherapy (docetaxel, paclitaxel or vinflunine) at the discretion of the investigator, as intravenous (i.v.) infusion once every three weeks (on day 1 of a 21-day cycle).
Arm/Group | Rogaratinib (BAY1163877) | Chemotherapy
Number analyzed (Participants) | 86 | 82
Participants
  Any TEAE | 86 | 82
  Any drug related TEAE | 81 | 76

ADVERSE EVENTS:
Time Frame: Approximately 29 months
Description: A treatment-emergent adverse event reported in this study was defined as any event arising or worsening after the start of study drug administration until 30 days after the last administration of study treatment.
Arm/Group | Rogaratinib (BAY1163877) | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 47/86 | 45/82
Serious Adverse Events (participants affected / at risk) | 39/86 | 33/82
Other Adverse Events (participants affected / at risk) | 85/86 | 77/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib (BAY1163877) (N=86) | Chemotherapy (N=82)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 4 (6) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Relapsing fever (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Groin infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Biopsy liver (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (7) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rogaratinib (BAY1163877) (N=86) | Chemotherapy (N=82)
Anaemia (Blood and lymphatic system disorders) | 11 (17) | 28 (66)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 19 (30)
Dry eye (Eye disorders) | 5 (5) | 3 (3)
Detachment of retinal pigment epithelium (Eye disorders) | 7 (16) | 0 (0)
Subretinal fluid (Eye disorders) | 7 (8) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (18) | 13 (27)
Constipation (Gastrointestinal disorders) | 25 (31) | 29 (54)
Diarrhoea (Gastrointestinal disorders) | 48 (92) | 18 (19)
Dry mouth (Gastrointestinal disorders) | 10 (15) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 5 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 27 (38) | 20 (38)
Stomatitis (Gastrointestinal disorders) | 10 (15) | 10 (14)
Vomiting (Gastrointestinal disorders) | 15 (19) | 18 (26)
Asthenia (General disorders) | 25 (52) | 19 (40)
Fatigue (General disorders) | 21 (32) | 28 (41)
Mucosal inflammation (General disorders) | 7 (20) | 8 (12)
Oedema peripheral (General disorders) | 8 (9) | 10 (13)
Pyrexia (General disorders) | 12 (15) | 10 (14)
Conjunctivitis (Infections and infestations) | 5 (8) | 3 (3)
Influenza (Infections and infestations) | 5 (5) | 0 (0)
Paronychia (Infections and infestations) | 7 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 8 (13)
Alanine aminotransferase increased (Investigations) | 13 (22) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 10 (16) | 2 (3)
Blood creatinine increased (Investigations) | 11 (18) | 3 (6)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 0 (0)
Lipase increased (Investigations) | 9 (25) | 3 (11)
Neutrophil count decreased (Investigations) | 0 (0) | 14 (22)
Weight decreased (Investigations) | 10 (11) | 6 (7)
White blood cell count decreased (Investigations) | 0 (0) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 12 (14) | 2 (3)
Calcium phosphate product increased (Investigations) | 8 (10) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (11) | 6 (14)
Hyperphosphataemia (Metabolism and nutrition disorders) | 39 (79) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (9) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 36 (55) | 21 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (4)
Dysgeusia (Nervous system disorders) | 13 (14) | 5 (6)
Headache (Nervous system disorders) | 6 (7) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 3 (4) | 10 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 10 (14)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4)
Haematuria (Renal and urinary disorders) | 9 (13) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (23) | 24 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (10) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 3 (5)
Onychomadesis (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 7 (12) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03410693/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03410693/SAP_001.pdf